CLINICAL TRIAL: NCT03698786
Title: Exercise Effects on Appetite-regulating Hormones and Cardiovascular Risk Factors in South Asian and White European Men
Brief Title: Exercise Effects on Appetite-regulating Hormones and Cardiovascular Risk Factors
Status: Completed | Type: Observational
Sponsor: Kingston University (Other)
Responsible Party: Principal Investigator, Hannah Moir, Senior Lecturer in Health & Exercise Prescription, Kingston University
Other Study IDs: KingstonUSport2
Record Dates: First submitted 2018-09-27; First posted 2018-10-09 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Risk Factor, Cardiovascular; Physical Activity; Pre-diabetes
MeSH Terms: conditions — Motor Activity; Glucose Intolerance | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma and serum stored according to Human Tissue Act for maximum of 6 years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- European males: This study will involve a cohort of 15 White European men, between the ages of 18-50 years. Participants will be non-smokers, not dieting, and physically well to participate.
  Participants will be required to exercise on one occasion.
  Interventions: Behavioral: Exercise
- South Asian males: This study will involve a cohort of 15 South Asian (India, Pakistan, Sri Lanka, Nepal, Bangladesh, Maldives and Bhutan), men, between the ages of 18-50 years. Participants will be non-smokers, not dieting, and physically well to participate.
  Participants will be required to exercise on one occasion.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Participants will be required to complete two, 8-hours trials (exercise & control) in a randomised order, preceded by 2 hours of preliminary testing (baseline) with no more than 14 days between conditions.

SUMMARY:
The aim of this study is to examine the effect of a single bout of moderate exercise, standardized breakfast and buffet meal on appetite-related hormones, type two diabetes and cardiovascular risk factors with a comparison between healthy South Asian and white European men. It is of interest to see if any factor differences occur in appetite-regulating hormones and cardiovascular disease risk factors whilst exercising. If so strategies may be used to alter regulation in diet and exercise to reduce risk cardiovascular disease as this is the number one cause of death globally.

DETAILED DESCRIPTION:
Cardiovascular diseases are recognised as the number one cause of death globally. Furthermore, diabetes is a major risk factor for cardiovascular disorders with abundant evidence showing that patients with type 2 diabetes (T2D) are at higher risk of cardiovascular disease (CVD) than those with a normal glycaemia.

In contrast to the declining numbers in the Western world, the prevalence of CVD and T2D is growing in low - and middle - income countries accompanied by a rapid increase of mortality and morbidity. Of interest, a rise in CVD prevalence has been particularly observed in people of South Asian origin including India, Bangladesh, Pakistan, Sri Lanka or Nepal with a projection showing that in this population deaths attributed to CVD will rise globally to nearly 36 % in 2030 compared to 29 % in 2005. South Asians collectively form 20% of the global population while in the UK they are the largest ethnic minority group representing over 5% of the total UK population .

Although the majority of research has been conducted mainly on White individuals, recent studies have revealed that traditional CVD risk factors such as hypertension, dyslipidaemia, insulin resistance and diabetes are higher in South Asians than other ethnicities. The factors underlying the high CVD risk in this population remain largely unexplained even though genetic predisposition and physical inactivity could play a key role. In contrast to European counterparts, sedentary lifestyles or physical inactivity have been identified as an important coronary heart disease (CHD) risk factor in South Asians. A systematic review from the United Kingdom (U.K.) showed that South Asians are participating in up to 50-75% less physical activity compared to their European counterparts.

In addition to the traditional risk factors there are emerging biomarkers which could represent meaningful predictors of metabolic disorders and related complications. Specifically, appetite hormones secreted mainly by the gastrointestinal tract, such as Acylated Ghrelin or Peptide YY (PYY) have shown potential effects on glucose homeostasis and cardiovascular system. Current experimental studies suggest beneficial cardiovascular, anti-inflammatory and anti-apoptotic effects of ghrelin in the cardiovascular system.

Although evidence suggests that ghrelin may be a potential metabolic risk factor and is important in appetite regulation, no studies to the researcher's knowledge have examined changes of this peptide in South Asians despite the fact that CVD and T2D burden in the South Asian population is growing. Likewise, although studies have investigated the effects of exercise on ghrelin and other appetite hormones, no study has taken in consideration the effects of exercise on appetite gut hormones in South Asian populations.

Therefore, this research project aims to examine specific appetite hormones in response to a single bout of exercise, standardised meal and ad libitum buffet meal, with a comparison between South Asians and White Europeans identifying potential relationships with genetic and other metabolic risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker
* Non-dieting
* Physically well to participant in maximal exercise
* Male
* Not taking any anticoagulant or anti-inflammatory medication
* Between the ages 18-50
* White European or South Asian

Exclusion Criteria:

* Those that are taking any anticoagulant or anti-inflammatory medication
* Those with a known medical condition such as diabetes, cardiovascular disease.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will involve a cohort of 15 White European and 15 South Asian (India, Pakistan, Sri Lanka, Nepal, Bangladesh, Maldives and Bhutan), men, between the ages of 18-50 years with no known underlying disease.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2018-12-23 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Plasma Acylated ghrelin concentration | 2 days
  Plasma acylated ghrelin will be examined before and after the standardised breakfast, libitum buffet meal and exercise and before leaving the laboratory (please refer to study design for details). Commercially available enzyme-linked immunosorbent assays (Bertin Bioreagent, Montigny le Bretonneux, France) will be used to measure plasma acylated ghrelin concentration. The sample will be collected from whole blood using venepuncture.

SECONDARY OUTCOMES:
Plasma TAG concentration | 2 days
  Plasma Insulin will be also examined before and after the standardised breakfast, libitum buffet meal and exercise and before leaving the laboratory (please refer to study design for details). Commercially available enzyme-linked immunosorbent assays (Mercodia, Uppsala, Sweden) will be used to measure plasma Insulin concentration. The sample will be collected from whole blood using venepuncture.
Plasma triacylglycerol (TAG) concentration | 2 days
  Plasma TAG concentration will be determined before and after the standardised breakfast, libitum buffet meal and exercise and before leaving the laboratory (please refer to study design for details) by enzymatic, colorimetric methods using a bench top analyser (Pentra 400; HORIBA ABX Diagnostics, Montpellier, France). The sample will be collected from whole blood using venepuncture.
Plasma high-density lipoprotein (HDL) cholesterol concentration | 2 days
  Plasma HDL concentration will be determined before and after the standardised breakfast, libitum buffet meal and exercise and before leaving the laboratory (please refer to study design for details) by enzymatic, colorimetric methods using a bench top analyser (Pentra 400; HORIBA ABX Diagnostics, Montpellier, France). The sample will be collected from whole blood using venepuncture.
Cardiorespiratory fitness | 2 days
  Cardiorespiratory fitness will be determined during the preliminary test (please refer to study design for details) using an incremental exercise test to volitional exhaustion on an electromagnetically braked cycle ergometer (Lode Excalibur Sport, Groningen, Netherlands). Participants will cycle at a self-selected pedal rate between 70 to 90 revolutions per minute for 3 min at 80 watts (warm up), followed by increments of 30 watts every 3 minutes until volitional fatigue. The sample will be collected from whole blood using venepuncture.
Plasma Glucose concentration for impaired glucose tolerance (IGT) | 2 days
  Plasma glucose concentration will be determined before and after the standardised breakfast, libitum buffet meal and exercise and before leaving the laboratory (please refer to study design for details) by enzymatic, colorimetric methods using a bench top analyser (Pentra 400; HORIBA ABX Diagnostics, Montpellier, France). The sample will be collected from whole blood using venepuncture.
Plasma Peptide YY concentration | 2 days
  Plasma PYY will be also examined before and after the standardised breakfast, libitum buffet meal and exercise and before leaving the laboratory (please refer to study design for details). Commercially available enzyme-linked immunosorbent assays (Millipore, Billerica, USA) will be used to measure plasma PYY concentration. The sample will be collected from whole blood using venepuncture.
Plasma Leptin concentration | 2 days
  Plasma leptin will be also examined before and after the standardised breakfast, libitum buffet meal and exercise and before leaving the laboratory (please refer to study design for details). Commercially available enzyme-linked immunosorbent assays (Millipore, Billerica, USA) will be used to measure plasma leptin concentration. The sample will be collected from whole blood using venepuncture.

CONTACTS AND LOCATIONS:
Overall Officials: Juliet Juliet, Study Chair — Kingston University
Locations (1):
- Applied & Human Sciences Human Performance Lab, Kingston upon Thames, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gijsberts CM, den Ruijter HM, Asselbergs FW, Chan MY, de Kleijn DP, Hoefer IE. Biomarkers of Coronary Artery Disease Differ Between Asians and Caucasians in the General Population. Glob Heart. 2015 Dec;10(4):301-311.e11. doi: 10.1016/j.gheart.2014.11.004. Epub 2015 Mar 7. PMID 26014657
- [Background] Gujral UP, Pradeepa R, Weber MB, Narayan KM, Mohan V. Type 2 diabetes in South Asians: similarities and differences with white Caucasian and other populations. Ann N Y Acad Sci. 2013 Apr;1281(1):51-63. doi: 10.1111/j.1749-6632.2012.06838.x. Epub 2013 Jan 14. PMID 23317344
- [Background] Huang Y, Cai X, Mai W, Li M, Hu Y. Association between prediabetes and risk of cardiovascular disease and all cause mortality: systematic review and meta-analysis. BMJ. 2016 Nov 23;355:i5953. doi: 10.1136/bmj.i5953. PMID 27881363
- [Background] Wulan SN, Westerterp KR, Plasqui G. Metabolic profile before and after short-term overfeeding with a high-fat diet: a comparison between South Asian and White men. Br J Nutr. 2014 May 28;111(10):1853-61. doi: 10.1017/S0007114514000014. Epub 2014 Feb 10. PMID 24506887
- [Background] Bailey DP, Smith LR, Chrismas BC, Taylor L, Stensel DJ, Deighton K, Douglas JA, Kerr CJ. Appetite and gut hormone responses to moderate-intensity continuous exercise versus high-intensity interval exercise, in normoxic and hypoxic conditions. Appetite. 2015 Jun;89:237-45. doi: 10.1016/j.appet.2015.02.019. Epub 2015 Feb 17. PMID 25700630
- [Background] Deighton K, Barry R, Connon CE, Stensel DJ. Appetite, gut hormone and energy intake responses to low volume sprint interval and traditional endurance exercise. Eur J Appl Physiol. 2013 May;113(5):1147-56. doi: 10.1007/s00421-012-2535-1. Epub 2012 Oct 31. PMID 23111564
- [Background] Gholap N, Davies M, Patel K, Sattar N, Khunti K. Type 2 diabetes and cardiovascular disease in South Asians. Prim Care Diabetes. 2011 Apr;5(1):45-56. doi: 10.1016/j.pcd.2010.08.002. Epub 2010 Sep 25. PMID 20869934
- [Background] King JA, Garnham JO, Jackson AP, Kelly BM, Xenophontos S, Nimmo MA. Appetite-regulatory hormone responses on the day following a prolonged bout of moderate-intensity exercise. Physiol Behav. 2015 Mar 15;141:23-31. doi: 10.1016/j.physbeh.2014.12.050. Epub 2015 Jan 3. PMID 25562575

DOCUMENTS (2):
  • Study Protocol (2017-05-05): https://cdn.clinicaltrials.gov/large-docs/86/NCT03698786/Prot_000.pdf
  • Informed Consent Form (2017-05-05): https://cdn.clinicaltrials.gov/large-docs/86/NCT03698786/ICF_001.pdf